CLINICAL TRIAL: NCT00520117
Title: Assessing the Psychosocial Burden in Women With an Abnormal Pap Results After Screening Interventions
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor, Mahidol University
Other Study IDs: 2007-024
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Papanicolaou Smear

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- negative pap-smear
- positive pap-smear

SUMMARY:
The primary purpose of this study is to assess the psychosocial burden in women who have experienced an abnormal pap results after screening interventions.

DETAILED DESCRIPTION:
This study will be a Thailand, clinic-based, cross-sectional, questionnaire study. Approximately 151 female participants will be enrolled. Study staff will interview the subject to collect basis demographic data and self reported medical history. And the subjects will be given the questionnaire packet for self-administration. After subjects complete the packet, study staff will review the questionnaires for completeness prior to the study subject leaving the clinic.

ELIGIBILITY:
Inclusion Criteria:

* female, between 18 and 45 years of age and must have recently experienced an abnormal pap results within the past 3 months.

Exclusion Criteria:

* has any condition which in the opinion of the investigator might interfere with the evaluation of the study objectives
* has other concurrent/active STD's
* has a history of known prior vaccination with an HPV vaccine
* has a history of recent (within 1 year from date of enrollment) or ongoing alcohol abuse or other drug abuse.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients having pap-smear at Ratchawithi Hospital
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
psychological burden of women with abnormal pap-smear | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, Professor, Principal Investigator — Department of Clinical ITropical Medicine, Faculty of Tropical Medicine, Mahidol University
Locations (1):
- Clinical Infectious Diseases Research Unit, Bangkok, Thailand